CLINICAL TRIAL: NCT02643784
Title: Exploratory Study on the Effects of Early Rosuvastatin Treatment in Patients With Acute Ischemic Stroke
Acronym: AIS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ESR-14-10028
Record Dates: First submitted 2015-12-16; First posted 2015-12-31 (Estimated); Last update posted 2015-12-31 (Estimated); Status verified 2015-12

CONDITIONS: Ischemic
Keywords: acute ischemic stroke
MeSH Terms: conditions — Ischemia; Ischemic Stroke | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rosuvastatin (Experimental): Rosuvastatin study drug will be supplied in tablets (10 mg), assigned dose to be taken orally, once daily by subjects randomized to receive rosuvastatin 20 mg(take rosuvastatin until 14th day).
  Interventions: Drug: Rosuvastatin; Other: Control
- Control (No Intervention): Control group(don't take rosuvastatin until 14th day), as directed by the study physician.

INTERVENTIONS:
Drug: Rosuvastatin — Randomized Treatment Period (Day 1 through Day 14): 20 mg once daily for 14 days.
  Follow up Period (Day 15 through Day 90) Subjects in both groups who enter the follow up period will receive rosuvastatin 10mg/day.
  Other Names: RSV
  Arms: Rosuvastatin
Other: Control — Randomized Treatment Period (Day 1 through Day 14):
  No treatment of rosuvastatin for control group. Follow up Period (Day 15 through Day 90) Subjects in both groups who enter the follow up period will receive rosuvastatin 10mg/day.
  Arms: Rosuvastatin

SUMMARY:
This is an exploratory, randomized, open-label, 2-arm, parallel-group study exploring the efficacy of rosuvastatin (20mg/day) in patients with acute ischemic stroke.

DETAILED DESCRIPTION:
This is a 90-day, explanatory; randomized; open-label, 2-arm; parallel group with blinded outcome evaluation study exploring the efficacy and study of early rosuvastatin 20 mg/d treatment in acute ischemic patients with stroke onset in 24 hours.

ELIGIBILITY:
Inclusion Criteria:

1. 45 to 75 years old patients;
2. Stroke involving the vascular territory of the middle cerebral artery (MCA) as judged by clinical and MRI evidences;
3. Time from symptom onset to take the study assigned medication is within 24 hours;
4. Statin naïve or discontinued at least 3 month before stroke onset;
5. First ever stroke or mild sequelae (with modified Rankin Score 0-1) before the index event;
6. Moderate neurological deficit with baseline NIHSS scoring from 4-20;
7. MRI scans （T1W1、T2W2、T2Flair、DWI、SWI）accomplished from 12 to 48 hours after the onset;
8. Consent form signed.

Exclusion Criteria:

-

Any of the following is regarded as a criterion for exclusion from the study:

1. Stroke involving the vascular territory of the vertebrobasilar artery as judged by clinical and MRI evidences;
2. Hemorrhagic transformation or intracranial hemorrhage on baseline MRI. MRI performed between 12-48 hours after the onset, if MRI provides evidences which met with the exclusion criteria, the patients will be excluded from the study;
3. Any circumstances under which MRI scans can't be performed;
4. Evidences suggesting cardiogenic stroke such as atrial fibrillation, acute coronary syndrome, patent foramen ovale , etc;
5. Comatose with NIHSS 1a>1;
6. Medical or psychiatric conditions such as severe hepatic or renal dysfunction, heart failure, malignancy, major depression, dementia, alcohol or drug abuse;
7. Suitable for rt-Plasminogen Activator thrombolysis treatment;
8. Receiving medication with possible neuroprotective functions after stroke onset;
9. Currently take steroids therapy;
10. Diagnosed with malignancy within 5 years;
11. Patients with myopathy or serum creatine kinase > 3 times the upper limit of normal not caused by myocardial injury;
12. Severe renal function damage (eGFR<30);
13. Concurrent use ciclosporin;
14. A history of hypersensitivity of statins and other severe complication;
15. Child-bearing women ;
16. Patients who are or may be pregnant;
17. Other conditions under which patients not pertinent to attend the study as judged by the investigators.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-12; Primary Completion 2017-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Percent changes in infarction volumes measured by MRI on the 14th day compared with the baseline of the stroke | 0-14d

SECONDARY OUTCOMES:
Absolute changes in infarction volumes measured by MRI on the 14th day compared with the baseline of the stroke | 0-14d
Proportion of patients whose infarction volume reduced on the 14th day compared with the baseline of the stroke | 0-14d
The neurological outcomes measured by NIHSS (14,90 days), compared between statin group and standard group | 14-90d
The functional outcome measured by modified Rankin Scale (14,90 days), compared between statin group and standard group | 14-90d
The rate of the new-onset infarct assessed by MRI from baseline to 14th day, compared between statin group and standard group | 0-14d

IPD SHARING:
Plan to Share IPD: Yes